CLINICAL TRIAL: NCT04589091
Title: Corneal Topography Asymmetry Indices Changes After Corneal Refractive Surgery
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Dina Tadros, Lecturer of ophthalmology , Tanta University Hospital, Tanta University
Other Study IDs: 34081/9/20
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Refractive Surgical Procedures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group(1): Patient who underwent PRK
  Interventions: Other: Refractive surgery
- Group(2): Patient underwent LASIK
  Interventions: Other: Refractive surgery

INTERVENTIONS:
Other: Refractive surgery — Refractive surgery for correction of error of refraction

SUMMARY:
To evaluate the changes that occur in the corneal indices after corneal refractive surgery either PRK or LASIK.

DETAILED DESCRIPTION:
Retrospectively review the medical records of all patients who underwent refractive surgery referred from the out-patient clinic of Tanta University hospital between September 2015 and September 2020 .

Data collection will include:

Preoperative and postoperative Evaluation: Age, sex, uncorrected distance visual acuity (UDVA), corrected distance visual acuity (CDVA), manifest and cycloplegic refraction, Slit lamp biomicroscopy, fundus examination.

Data of Corneal Tomography keratometric using Scheimpflug camera (Pentacam Oculus- Germany) :that includes the following indices

1. Average keratometric value (K mean) in diopters
2. Maximum simulated keratometry (Kmax) in diopters
3. Index of Surface Variance (ISV) in microns
4. Index of Vertical Asymmetey (IVA) in microns
5. Radii Minimum (R min) in microns
6. Index of height asymmetry (IHA) in microns
7. Index of height decantation (IHD) in microns
8. Aberration coefficient (ABR)

The data of the pentacam will be collected pre-operative and analyzed at 1 month, 3 months and 6 months with recording of the complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent refractive surgery either PRK, LASIK with age between 19 and 35 years old

Exclusion Criteria:

* Kertoconus.

  * Corneal scarring.
  * Previous corneal infections.
  * Minimum corneal thickness at the thinnest location less than 400 µm.
  * History of uveitis or ocular allergy.
  * Pre-existing glaucoma.
  * Data not available

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: We will retrospectively review the medical records of all patients who underwent refractive surgery referred from the out-patient clinic of Tanta University hospital between September 2015 and September 2020
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the changes that occur in the corneal indices after corneal refractive surgery either PRK or LASIK. | 6 months
  Using the results of measurements of Scheimpflug camera (Pentacam Oculus- Germany) :that includes the following indices
  1. Average keratometric value (K mean) in diopters
  2. Maximum simulated keratometry (Kmax) in diopters
  3. Index of Surface Variance (ISV) in microns
  4. Index of Vertical Asymmetey (IVA) in microns
  5. Radii Minimum (R min) in microns
  6. Index of height asymmetry (IHA) in microns
  7. Index of height decantation (IHD) in microns
  8. Aberration coefficient (ABR)
  The numbers from preoperative records will be compared with postoperative records after the refractive surgery is done . All the values will be expressed as mean ± standard deviation and the data will be analyzed as 1 months, 3 months and 6 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospital, Tanta, El-Garbeia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 3 months
Access Criteria: Link

REFERENCES:
- [Result] Bailey MD, Zadnik K. Outcomes of LASIK for myopia with FDA-approved lasers. Cornea. 2007 Apr;26(3):246-54. doi: 10.1097/ICO.0b013e318033dbf0. PMID 17413947
- [Result] Sridhar MS, Rao SK, Vajpayee RB, Aasuri MK, Hannush S, Sinha R. Complications of laser-in-situ-keratomileusis. Indian J Ophthalmol. 2002 Dec;50(4):265-82. PMID 12532491
- [Result] Mohammadi SF, Nabovati P, Mirzajani A, Ashrafi E, Vakilian B. Risk factors of regression and undercorrection in photorefractive keratectomy: a case-control study. Int J Ophthalmol. 2015 Oct 18;8(5):933-7. doi: 10.3980/j.issn.2222-3959.2015.05.14. eCollection 2015. PMID 26558204
- [Result] Belin MW, Ambrosio R Jr. Corneal ectasia risk score: statistical validity and clinical relevance. J Refract Surg. 2010 Apr;26(4):238-40. doi: 10.3928/1081597X-20100318-01. No abstract available. PMID 20415320